CLINICAL TRIAL: NCT01707082
Title: A Phase 1, Randomized, Placebo-Controlled, Multiple Dose Study To Evaluate The Safety, Pharmacokinetics And Pharmacodynamics Of PF-06282999 In Healthy Overweight Subjects And A Fixed-Sequence Study To Assess The Effect Of PF-06282999 On The Pharmacokinetics Of Midazolam In Healthy Subjects
Brief Title: A Study To Test The Safety, Amount And Effects Of PF-06282999 In Healthy Overweight Adults And A Study To Test The Effects Of PF-06282999 On The Amount Of The Approved Drug, Midazolam, In Healthy Adults
Acronym: B521MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B5211002
Record Dates: First submitted 2012-10-03; First posted 2012-10-15 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
MeSH Terms: interventions — 2-(6-(5-chloro-2-methoxyphenyl)-4-oxo-2-thioxo-3,4-dihydropyrimidin-1(2H)-yl)acetamide; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part A Cohort 1 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo
- Part A Cohort 2 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo
- Part A Cohort 3 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo
- Part A Cohort 4 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo
- Part A Cohort 5 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo
- Part B Cohort 1 (Experimental)
  Interventions: Drug: midazolam; Drug: PF-06282999
- Part B Cohort 2 (Experimental)
  Interventions: Drug: midazolam; Drug: PF-06282999

INTERVENTIONS:
Drug: PF-06282999 — Tablet, 10 mg, every 8 hours, 14 days
  Arms: Part A Cohort 1
Drug: Placebo — Tablet, 0 mg, every 8 hours, 14 days
  Arms: Part A Cohort 1
Drug: PF-06282999 — Tablet, 30 mg, every 8 hours, 14 days
  Arms: Part A Cohort 2
Drug: Placebo — Tablet, 0 mg, every 8 hours, 14 days
  Arms: Part A Cohort 2
Drug: PF-06282999 — Tablet, 100 mg, every 8 hours, 14 days
  Arms: Part A Cohort 3
Drug: Placebo — Tablet, 0 mg, every 8 hours, 14 days
  Arms: Part A Cohort 3
Drug: PF-06282999 — Tablet, 250 mg, every 8 hours, 14 days
  Arms: Part A Cohort 4
Drug: Placebo — Tablet, 0 mg, every 8 hours, 14 days
  Arms: Part A Cohort 4
Drug: PF-06282999 — Tablet, 350 mg every 8 hours or 500 mg every 12 hours, 14 days
  Arms: Part A Cohort 5
Drug: Placebo — Tablet, 0 mg, every 8 or 12 hours, 14 days
  Arms: Part A Cohort 5
Drug: midazolam — Tablet, 7.5 mg, single dose on Period 1 Day 1 and Period 2 Day 14
  Arms: Part B Cohort 1
Drug: PF-06282999 — Tablet, dose to be determined (determined in Part A), every 8 or 12 hours, 14 days
  Arms: Part B Cohort 1
Drug: midazolam — Tablet, 7.5 mg, single dose on Period 1 Day 1 and Period 2 Day 14
  Arms: Part B Cohort 2
Drug: PF-06282999 — Tablet, dose to be determined (determined in Part A), every 8 or 12 hours, 14 days
  Arms: Part B Cohort 2

SUMMARY:
Part A of the study will test the safety, the amount of drug in the body, and effects of the drug in the body after multiple doses. This will be conducted in healthy overweight adults. Part B of the study will test the effects of multiple doses of the investigational drug on the amount of midazolam, an approved drug, in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests). Women must be of non childbearing potential.
* Body Mass Index (BMI) of 27.0 to 35.0 kg/m2 (Part A) or 17.5 to 30.5 kg/m2 (Part B); and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including clinically significant drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject with any contraindication to midazolam according to the country specific labeling or subject with previous intolerance or allergy to benzodiazepines (applicable to Part B of study only).
* Subjects who were enrolled in Part A are excluded from participation in Part B of this study.
* Subjects who have previously participated in a study with PF-06282999.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Pre-dose,0.5,1,2,3,4,5,6,7,8 and 16 hrs post morning dose Day 1 Part A
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Pre-dose,0.5,1,2,3,4,5,6,7,8 and 16 hrs post morning dose Day 1 Part A
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | Pre-dose,0.5,1,2,3,4,5,6,7,8 and 16 hrs post morning dose Day 1 Part A
Apparent Oral Clearance (CL/F) | Pre-dose,0.5,1,2,3,4,5,6,7,8 and 16 hrs post morning dose Day 1 Part A
Maximum Observed Plasma Concentration (Cmax) | Pre-dose,0.5,1,2,3,4,5,6,7,8,10,12,16,24,36, and 48 hrs post morning dose Day 14 Part A
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Pre-dose,0.5,1,2,3,4,5,6,7,8,10,12,16,24,36, and 48 hrs post morning dose Day 14 Part A
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | Pre-dose,0.5,1,2,3,4,5,6,7,8,10,12,16,24,36, and 48 hrs post morning dose Day 14 Part A
Minimum Observed Plasma Trough Concentration (Cmin) | Pre-dose,0.5,1,2,3,4,5,6,7,8,10,12,16,24,36, and 48 hrs post morning dose Day 14 Part A
Apparent Oral Clearance (CL/F) | Pre-dose,0.5,1,2,3,4,5,6,7,8,10,12,16,24,36, and 48 hrs post morning dose Day 14 Part A
Plasma Decay Half-Life (t1/2) | Pre-dose,0.5,1,2,3,4,5,6,7,8,10,12,16,24,36, and 48 hrs post morning dose Day 14 Part A
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Pre-dose,0.5,1,2,3,4,5,6,8,10,12 and 16 hrs post dose Day 1 Period 1 Part B
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) Midazolam
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | -2,-1.5,-1,Pre-dose,1,2,4,6,8,10,14 Day 14 Period 2 Part B
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) Midazolam
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | Pre-dose,0.5,1,2,3,4,5,6,8,10,12 and 16 hrs post dose Day 1 Period 1 Part B
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8). Midazolam
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | -2,-1.5,-1,Pre-dose,1,2,4,6,8,10,14 Day 14 Period 2 Part B
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8). Midazolam
Maximum Observed Plasma Concentration (Cmax) | Pre-dose,0.5,1,2,3,4,5,6,8,10,12 and 16 hrs post dose Day 1 Period 1 Part B
Maximum Observed Plasma Concentration (Cmax) | -2,-1.5,-1,Pre-dose,1,2,4,6,8,10,14 Day 14 Period 2 Part B
Average Concentration (Cav) | Pre-dose,0.5,1,2,3,4,5,6,7,8,10,12,16,24,36, and 48 hrs post morning dose Day 14 Part A
Accumulation Ratio | Pre-dose,0.5,1,2,3,4,5,6,7,8,10,12,16,24,36, and 48 hrs post morning dose Day 14 Part A

SECONDARY OUTCOMES:
Diastolic Blood Pressure | Day 1 Pre-dose,1,2,4,8,12 and 16 hrs post dose Part A
  Mean 24-hour average diastolic blood pressure
Diastolic Blood Pressure | Day 13 Pre-dose,1,2,4,8,12 and 16 hrs post dose Part A
  Mean 24-hour average diastolic blood pressure
Systolic Blood Pressure | Day 1 Pre-dose,1,2,4,8,12 and 16 hrs post dose Part A
  Mean 24-hour average systolic blood pressure
Systolic Blood Pressure | Day 13 Pre-dose,1,2,4,8,12 and 16 hrs post dose Part A
  Mean 24-hour average systolic blood pressure
interleukin-6 | Days 1 and 14 pre-dose Part A
high-sensitivity C-reactive protein | Days 1 and 14 pre-dose Part A
total cholesterol, HDL-C, triglycerides and calculated LDL-C | Days 1 and 14 pre-dose Part A
ApoBTotal,ApoB48, ApoB100, ApoA-1 | Days 1 and 14 pre-dose Part A
Diastolic Blood Pressure | Day 1 Pre-dose,1,2,4,8,12 and 16 hrs post dose Part B
  Mean 24-hour average diastolic blood pressure
Diastolic Blood Pressure | Day 13 Pre-dose,1,2,4,8,12 and 16 hrs post dose Part B
  Mean 24-hour average diastolic blood pressure
Systolic Blood Pressure | Day 1 Pre-dose,1,2,4,8,12 and 16 hrs post dose Part B
  Mean 24-hour average systolic blood pressure
Systolic Blood Pressure | Day 13 Pre-dose,1,2,4,8,12 and 16 hrs post dose Part B
  Mean 24-hour average systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5211002&StudyName=A%20Study%20To%20Test%20The%20Safety%2C%20Amount%20And%20Effects%20Of%20PF-06282999%20In%20Healthy%20Overweight%20Adults%20And%20A%20Study%20To%20Test%20The%20Effects%20Of%20